CLINICAL TRIAL: NCT03989154
Title: Prospective Cohort Study for Primary Ovarian Insufficient Patients in Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD)
Brief Title: Primary Ovarian Insufficient Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-POI cohort study
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Healthy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prospective Cohort Study for Primary Ovarian Insufficient Patients was set up to investigate the short- and long-term health consequences in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, China.

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) is a rare cause of infertility in women affecting 1% of the population. It is characterized by amenorrhea, hypoestrogenism and elevated gonadotrophin levels in women younger than 40 years of age. Other than the reproductive outcome of these patients, the short- and long-term health consequences are still unknown.

Since last decade, Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD) has been used in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, and Henan Province Key Laboratory for Reproduction and Genetics. Information of patients (POI, PCOS, Endometriosis, azoospermia, ect) were recorded comprehensively. The current project plans to recruit POI participants in our center. Biological samples, questionnaires and short/long term health data will be collected. The study is aimed to provide evidence for POI prognosis.

ELIGIBILITY:
Inclusion Criteria:

* younger than 40 years of age
* at least four or more months of amenorrhea, two or more instances in which the serum FSH level is > 40 U/L (i.e., two inspections at intervals of 1 month or more), with an oestradiol level of <20pg/ml

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: (1) younger than 40 years of age; (2) at least four or more months of amenorrhea, two or more instances in which the serum FSH level is > 40 U/L (i.e., two inspections at intervals of 1 month or more), with an oestradiol level of <20pg/ml
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
FSH (Follicle stimulating hormone) | Change from Baseline FSH at each6 months
  mIU/mL
LH (luteinizing hormone) | Change from Baseline LH at each6 months
  mIU/mL
Estrogen | Change from Baseline Estrogen at each6 months
  pg/ml
Progesterone | Change from Baseline Progesterone at each6 months
  ng/ml

SECONDARY OUTCOMES:
Volume of uterus and ovary | Change from Baseline volume at each6 months
  Record the Length (mm)*Width (mm)*Height (mm) of uterus, and each ovary

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kovanci E, Schutt AK. Premature ovarian failure: clinical presentation and treatment. Obstet Gynecol Clin North Am. 2015 Mar;42(1):153-61. doi: 10.1016/j.ogc.2014.10.004. PMID 25681846
- [Background] Zhai J, Yao G, Dong F, Bu Z, Cheng Y, Sato Y, Hu L, Zhang Y, Wang J, Dai S, Li J, Sun J, Hsueh AJ, Kawamura K, Sun Y. In Vitro Activation of Follicles and Fresh Tissue Auto-transplantation in Primary Ovarian Insufficiency Patients. J Clin Endocrinol Metab. 2016 Nov;101(11):4405-4412. doi: 10.1210/jc.2016-1589. Epub 2016 Aug 29. PMID 27571179